CLINICAL TRIAL: NCT04507243
Title: Imaging-guided tDCS Therapy in Major Depression
Brief Title: Transcranial Direct Current Stimulation (tDCS) Therapy in Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Narr, Professor, Department of Neurology, Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-001544; R33MH110526 (NIH)
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial direct current stimulation; MRI; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Active and Sham controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active - HD tDCS (Experimental): Participants randomized to this arm will receive 12 sessions of high definition tDCS (HD-tDCS) stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex for 20-30 minutes.
  Interventions: Device: Active - HD tDCS
- Sham - HD tDCS (Sham Comparator): Participants randomized to this arm will receive 12 sessions of sham HD tDCS stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex for 20-30 minutes.
  Interventions: Device: Sham - HD tDCS

INTERVENTIONS:
Device: Active - HD tDCS — Non-invasive neuromodulation using HD electrodes placed on the scalp to deliver a constant, low current at 2 mA.
  Arms: Active - HD tDCS
Device: Sham - HD tDCS — Sham neuromodulation using HD electrodes placed on the scalp to deliver a low current ramped up/down for 20 sec.
  Arms: Sham - HD tDCS

SUMMARY:
Noninvasive transcranial direct current stimulation (tDCS) is a low-intensity neuromodulation technique of minimal risk that has been used as an experimental procedure for reducing depressive symptoms and symptoms of other brain disorders. Though tDCS applied to prefrontal brain areas is shown to reduce symptoms in some people with major depressive disorder (MDD), the extent of antidepressant response often differs. Methods that map current flow directly in the brain while a person is receiving tDCS and that determine how functional neuroimaging signal changes after a series of tDCS sessions may help us understand how tDCS works, how it can be optimized, and if it can be used as an effective antidepressant. Investigators will address these questions in a two-part randomized double blind exploratory clinical trial. For this part of the study, investigators will determine relationships between target engagement and clinical outcomes (mood) and functional sub-constructs of cognitive control and emotion negativity bias, and whether imaging markers at baseline predict changes in antidepressant response.

One hundred people with depression (50 in each group) will be randomized to receive either HD-tDCS or sham-tDCS for a total of 12 sessions each lasting 20 minutes occurring on consecutive weekdays. At the first and last session, subjects will receive 20-30 minutes of active or sham HD-tDCS in the MRI scanner, which will allow investigators to map tDCS currents, and track changes in regional cerebral blood flow (rCBF) pre-to- post treatment using completely non-invasive methods. At the first and last session and mid-way through the trial, participants will also complete a series of clinical ratings and neurocognitive tests.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS), a noninvasive neuromodulation technique, applied to the left dorsolateral prefrontal cortex (DLPFC) can reduce depressive symptoms and improve cognitive control in major depressive disorder (MDD). Such findings suggest modulation of top down prefrontal-limbic circuits, which are functionally distinct from ventro-limbic networks and include reciprocally connected DLPFC and dorsomedial anterior cingulate cortex (dACC). However, substantial variation in tDCS response is observed in MDD. This may be due to imprecise stimulation protocols and suboptimal engagement of the neural circuits mediating antidepressant response. Methods that optimize electrode placement and account for individual variation in anatomy and that map current flow directly in the brain may inform the mechanisms and potential clinical utility of tDCS. A new tDCS technique, high definition (HD) tDCS, offers more focal stimulation than conventional tDCS (C-tDCS). The degree to which C-tDCS or HD-tDCS engage dorsal prefrontal-limbic neural circuits is unknown, yet is vital for understanding, confirming and subsequently improving possible therapeutic effects. Innovative MRI techniques that are able to map tDCS currents in vivo and that track changes in regional cerebral blood flow occurring with tDCS over time can provide direct evidence of neural effects. Based on a) theoretical modeling of tDCS current flow, b) studies showing hypo-metabolism, decreased CBF or activity in dorsal prefrontal-limbic networks, c) modulation of these regions with treatment, and, c) our prior results showing significant relationships in between change in dACC rCBF and clinical response to electroconvulsive therapy (ECT), an established brain stimulation treatment, we will test for the tDCS engagement and modulation of the DLPFC and dACC using tDCS current mapping performed in vivo and perfusion MRI. MRI-guided neuronavigation will be used to optimize and standardize electrode placement for DLPFC stimulation.

In this trial, using HD-tDCS that optimal target engagement of DLPFC and larger rCBF changes in the DLPFC and dACC compared to C-tDCS in the first part of the trial, we will define relationships between target engagement and change in mood and behavior. Patients with moderate to severe MDD (N=100, n=50 in each group) will be randomized to Active or Sham left anodal DLPFC HD-tDCS. Patients will complete MRI scans including tDCS current mapping and pCASL as well as two functional imaging tasks probing cognitive control and emotion negativity bias, recruiting prefrontal-limbic circuitry, before and after completing a 12-day trial of 20-minute tDCS sessions.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent;
* Meet DSM-5 criteria for a moderate-to-severe MDE, with Hamilton Rating Scale for Depression (HAMD) score of ≥14 and <24;
* Treatment naïve or on a stable standard antidepressant regimen (including selective serotonin reuptake inhibitors (SSRIs), serotonin-noradrenaline reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MOAIs) or tricyclic's (TCAs)) with no change in treatment 6-weeks prior to and during the tDCS intervention;
* Live within traveling distance to the University of California, Los Angeles (UCLA);
* Must refrain from making drastic hair-style changes throughout duration of study

Exclusion Criteria:

* Non-English speaking;
* Schizophrenia Axis I disorder;
* Primary anxiety disorder;
* Bipolar I disorder and psychotic disorders;
* Any neurological condition or major illness, including seizure disorder;
* Diagnosis of dementia of any type;
* Co-morbid substance abuse in the last three months;
* Contraindications to MR scanning (including pregnancy);
* Contraindications to tDCS (e.g., skin disease or treatment causing irritation);
* Treatment-resistant depression, with a history of a major depressive episode lasting > 2 years or failure to 2 or more antidepressant trials in the current episode;
* Any neuromodulation therapy (e.g., ECT, rTMS, DBS, VNS, or tDCS) within the last 3 months;
* Active suicidality;
* Current or past (within the last 1-month) use of anticonvulsants, lithium, psychostimulants, or dexamphetamine;
* Current use of decongestants or other medication previously shown to interfere with cortical excitability;
* Currently receiving any form of Cognitive Behavioral Therapy, Dialectical Behavioral Therapy, or Acceptance and Commitment Therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Measured joint longitudinal change in rCBF and mood scores over the tDCS trial | 3 weeks
  Correlation between percent change in rCBF after the tDCS trial and percent change in depressive symptoms for active versus sham tDCS conditions

SECONDARY OUTCOMES:
Measured joint longitudinal change in regional brain activation and mood scores over the tDCS trial | 3 weeks
  Correlation between percent change in regional brain activation for tasks probing cognitive control and emotion and percent change depressive symptoms for active versus sham tDCS conditions
Measured magnetic fields and rCBF at baseline and change in mood scores over the tDCS trial | 3 weeks
  Correlation between variations in magnetic fields and rCBF at baseline and clinical outcomes at the end of the tDCS treatment trial

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Narr, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jog MA, Norris V, Pfeiffer P, Taraku B, Kozikowski S, Schneider J, Boucher M, Iacoboni M, Woods R, Narr K. Personalized High-Definition Transcranial Direct Current Stimulation for the Treatment of Depression: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2531189. doi: 10.1001/jamanetworkopen.2025.31189. PMID 40932717